CLINICAL TRIAL: NCT06575374
Title: Open Label Single Arm Pilot Trial of Letermovir for Cytomegalovirus Prophylaxis After Axicabtagene Ciloleucel Therapy
Brief Title: Single Arm Pilot Trial of Letermovir for CMV Prophy in CAR T Cell
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0828; NCI-2024-07402 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cell Therapy
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label Single arm: Letermovir (Experimental): Participants will be identified/recruited/screened from the Lymphoma and Stem Cell Transplantation and Cellular Therapy services at MD Anderson Cancer Center.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Given by mouth or intravenously

SUMMARY:
The goal of this clinical research study is to learn if a drug called Letermovir can help to prevent CMV reactivation.

DETAILED DESCRIPTION:
Primary Objective:

Estimate the probabilities at days d = +28 and +98 following CAR T cell infusion, among patients alive at the day of evaluation, of CMV reactivation in CMV seropositive patients receiving letermovir for CMV prophylaxis after standard of care (SOC) axicabtagene ciloleucel (AXI-CEL) therapy, using the cutoff CMV DNA qPCR > c for c = 400 and 1000 IU/mL to define CMV reactivation, for a total of four (d, c) combinations.

Secondary Objectives:

Estimate overall survival probabilities at days+28, +98, and +364 following CAR T cell infusion of CMV seropositive patients receiving letermovir for CMV prophylaxis after SOC AXI-CEL therapy.

Describe the tolerability of letermovir during the period of CMV prophylaxis after SOC AXI-CEL therapy in CMV seropositive patients at high risk for CMV reactivation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age.
2. Have an ECOG performance status of 0 or 1.
3. The participant must be scheduled for SOC AXI-CEL.
4. The participant must be seropositive for CMV (defined as having anti-CMV IgG antibodies)
5. Creatinine clearance > 10 mL/min
6. Child Pugh class A or B if liver disease is present.
7. Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately.
8. Participant must understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection not responding to treatment, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Female participants who are pregnant or breastfeeding.
3. Unwilling or unable to follow protocol requirements.
4. Planned to receive any other anti-CMV therapy such as high dose acyclovir (500 mg/m2/dose intravenously every 8 hours or 800 mg orally 4 times a day) or high dose valacyclovir (2 grams three to four times daily or 2 grams three times daily) for the prophylaxis of CMV reactivation. Acyclovir or valacyclovir at lower doses for the prevention of HSV and VZV are allowed.
5. Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug.
6. Evidence for CMV infection defined as any positive CMV DNA qPCR test within 1 week prior to starting letermovir.
7. Child Pugh class C liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: George Chen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org